CLINICAL TRIAL: NCT06404099
Title: RECOVER-SLEEP: A Platform Protocol for Evaluation of Interventions for Sleep Disturbances in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-SLEEP: Platform Protocol, Appendix_A (Hypersomnia)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00112484_A; OTA-21-015G (Other Grant/Funding Number: NIH Grant to RTI; RTI subcontracting with DCRI)
Record Dates: First submitted 2024-05-06; First posted 2024-05-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Long COVID; Long COVID-19; Hypersomnia
Keywords: PASC
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Disorders of Excessive Somnolence | interventions — Modafinil; solriamfetol

STUDY DESIGN:
Intervention Model Description: This platform protocol is designed to allocate participants into an intervention appendix based on their symptoms of sleep disturbance. Within the appendix, participants will be randomly assigned based on the appendix study design. Site investigators and personnel will be informed as to which study intervention appendix participants are assigned, but they will be blinded to whether participants are receiving the active study intervention or control, when possible. Similarly, participants will be blinded to active intervention or control, when possible. Randomization will be stratified by the study site; other stratification factors may be considered per appendix.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wake-promoting drug: Modafinil or solriamfetol (Active Comparator): Participants in Appendix A will be randomized to study drug or control. Participants who meet the eligibility criteria for modafinil will receive either active modafinil or the modafinil-matched control. If modafinil is contraindicated for any reason, participants will be assessed for their ability to take solriamfetol. If participants are eligible for solriamfetol, they will receive either active solriamfetol or the solriamfetol-matched control. If solriamfetol is contraindicated, participants will be excluded from Appendix A. Modafinil and solriamfetol will be analyzed as a single wake-promoting drug condition versus control. The intervention duration will be 10 weeks.
  Interventions: Drug: Modafinil; Drug: Solriamfetol
- Modafinil-matched placebo or solriamfetol-matched placebo (Placebo Comparator): Participants in Appendix A will be randomized to study drug or control. Participants who meet the eligibility criteria for modafinil will receive either active modafinil or the modafinil-matched control. If modafinil is contraindicated for any reason, participants will be assessed for their ability to take solriamfetol. If participants are eligible for solriamfetol, they will receive either active solriamfetol or the solriamfetol-matched control. If solriamfetol is contraindicated, participants will be excluded from Appendix A. Modafinil and solriamfetol will be analyzed as a single wake-promoting drug condition versus control. The intervention duration will be 10 weeks.
  Interventions: Drug: Modafinil Placebo; Drug: Solriamfetol Placebo

INTERVENTIONS:
Drug: Modafinil — Modafinil is used off-label based on supporting published evidence in major depressive disorder (antidepressant augmentation), multiple sclerosis-related fatigue, Parkinson disease-related excessive daytime sleepiness, and severe cancer-related fatigue (in patients receiving active treatment). Doses up to 400 mg/day, given as a singleMode dose, have been well tolerated, but there is no consistent evidence that this dose confers additional benefit beyond that of the 200 mg dose.
  Study drug administration will total 10 weeks.
  Arms: Wake-promoting drug: Modafinil or solriamfetol
Drug: Modafinil Placebo — The placebo will be tooled to look similar to the modafinil tablet, but it will not contain the active ingredient. Modafinil placebo dosing will follow the same titration scheme as modafinil treatment.
  Unblinded study personnel will manage modafinil and placebo disbursement to maintain blinding among participants and blinded study personnel, including site investigators.
  Arms: Modafinil-matched placebo or solriamfetol-matched placebo
Drug: Solriamfetol — The proposed doses and the schedule of dose escalation are consistent with currently approved FDA labeling for solriamfetol for other disorders of excessive daytime sleepiness.
  Solriamfetol dosing will total 10 weeks, including 3 weeks for titration and 7 weeks of maintenance. Solriamfetol will be given as a 75 mg tablet (1 or 2 per day) in the morning. The 3-week titration will be facilitated by phone calls between the study team and participants. Titrations in dose will be dependent upon participants' symptoms and tolerance to solriamfetol, with a goal of participants taking the highest dose permitted by symptoms. This dose will be used for the maintenance phase.
  Arms: Wake-promoting drug: Modafinil or solriamfetol
Drug: Solriamfetol Placebo — The placebo tablet will be tooled to look similar to the solriamfetol tablet, but it will not contain the active ingredient. Solriamfetol placebo dosing will follow the solriamfetol dosing scheme and goal.
  Unblinded study personnel will manage solriamfetol and placebo disbursement to maintain blinding among participants and blinded study personnel, including site investigators.
  Arms: Modafinil-matched placebo or solriamfetol-matched placebo

SUMMARY:
The platform protocol is designed to be flexible so that it is suitable for a range of study settings and intervention types. Therefore, the platform protocol provides a general protocol structure that can be shared by multiple interventions and allows comparative analysis across the interventions. For example, objectives, measures, and endpoints are generalized in the platform protocol, but intervention-specific features are detailed in separate appendices.

This platform protocol is a prospective, multi-center, multi-arm, randomized controlled platform trial evaluating potential interventions for PASC-mediated sleep disturbances. The hypothesis is that symptoms of sleep and circadian disorders that emerge in patients with PASC can be improved by phenotype-targeted interventions. Specific sleep and circadian disorders addressed in this protocol include sleep-related daytime impairment (referred to as hypersomnia) and complex PASC-related sleep disturbance (reflecting symptoms of insomnia and sleep-wake rhythm disturbance).

DETAILED DESCRIPTION:
Interventions will be added to the platform protocol as appendices. Each appendix will leverage all elements of the platform protocol, with additional elements described in the individual appendix.

After completing Baseline assessments, participants will be randomized to an intervention group, which is based on their sleep phenotype, or into a placebo/control group.

ELIGIBILITY:
Inclusion Criteria:

• See NCT06404086 for RECOVER-SLEEP: Platform Protocol level inclusion criteria which applies to this appendix

Exclusion Criteria:

• See NCT06404086 for RECOVER-SLEEP: Platform Protocol level exclusion criteria which applies to this appendix (or sub-study)

Additional Appendix A (Hypersomnia) Level Exclusion Criteria:

1. Self-reported sleep duration <6 hours per night
2. Poorly controlled hypertension (systolic blood pressure ≥140 or diastolic blood pressure ≥90 mmHg)
3. Moderate to severe hepatic impairment (ie, Child-Pugh class B or C)*
4. Known estimated glomerular filtration rate <30 mL/min/1.73 m2 and/or chronic dialysis*
5. Recent myocardial infarction (<1 year), unstable angina, serious cardiac arrhythmias, or other serious heart problems, at the discretion of the investigator
6. Current use of stimulant or wake-promoting medications, unless a washout is permitted
7. Regular use of prescribed hypnotics for sleep (≥3 times per week); washout period is permitted.

   * characterized by the screening labs: coagulation panel and CMP w/LFTs

MODAFINIL EXCLUSION CRITERIA

1. Modafinil can affect drug metabolism given its effect on enzymes such as CYP3A4 and CYP2C19. To assess for drug interactions, investigators should use the Lexicomp Drug Interactions System that is available at most institutions.

   o If the search yields "D" - Consider Modifying Therapy or "X" - Avoid Combination, then the ACTION is to exclude the potential participant.

   An important example of this is steroid hormonal contraceptives.
   * If the search yields "C" - Monitor Therapy, then discuss with site PIs on a case-by-case basis.
   * If the search yields "A" - No Known Interaction or "B" - No Action Needed, then proceed to screen/include the potential participant.
2. Known severe left ventricular hypertrophy, mitral valve prolapse

SOLRIAMFETOL EXCLUSION CRITERIA

1. Concurrent treatment with a monoamine oxidase inhibitor (MAOI) or use of an MAOI within the preceding 14 days
2. Current use of dopaminergic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in total score of the PROMIS 8a SRI to assess sleep-related impairment | Baseline, End of Intervention (Day 77)
  The PROMIS 8a SRI form includes a total of 8 items that ask participants to reflect on their sleep-related daytime impairment over the past 7 days with questions rated not at all to very much. T-Scores range from 0 to 100, with a score of 55 being 1 standard deviation above population mean. Higher scores indicate greater sleep-related impairment.

SECONDARY OUTCOMES:
Change in total score of the PROMIS 8b SD to assess sleep disturbance | Baseline, End of Intervention (Day 77)
  The PROMIS 8b SD form includes a total of 8 items that ask participants to reflect on their sleep over the past 7 days with one question rated very poor to very good and the remaining questions rated not at all to very much. T-Scores range from 0 to 100, with > 55 1 SD above population mean.
Change in PROMIS 10a Fatigue score | Baseline, End of Intervention (Day 77)
  The PROMIS 10a Fatigue is a 10-item questionnaire that assesses a participant's fatigue on a scale of 1 (not at all fatigued) to 5 (very much).
Change in an objective neurocognitive battery score | Baseline, End of Intervention (Day 77)
Change in ECog2 measure | Baseline, End of Intervention (Day 77)
  Everyday Cognition 2 (ECog2) is a self-report, 41-item questionnaire used to measure measure the participant's perceived capacity to perform activities related to cognitive function, which could impact major activities of daily living and independence. It has been used for patients with mild cognitive impairment, Alzheimer's Disease, and dementia. It takes 5 minutes to complete.
Change in PASC Symptom Questionnaire responses | Baseline, End of Intervention (Day 77)
  Participants will be asked to complete a questionnaire that asks about the presence of PASC symptoms at Baseline and at follow-up visits. This questionnaire includes symptoms that have been associated with PASC.
Change in total score on the Insomnia Severity Index (ISI) | Baseline, End of Intervention (Day 77)
  The ISI is a 7-item, self-report questionnaire that assesses the nature, severity, and impact of insomnia, on a 5-point Likert scale (eg, 0 = not at all, 4 = extremely; scores: from 0 to 28). The ISI asks patients to recall their insomnia symptoms over the past 2 weeks.
Change in within-person variability (over a 7-day period) in sleep onset time, assessed by sleep diary | Baseline, End of Intervention (Day 77)
  Sleep onset time will be assessed by sleep diary
Change in average (over a 7-day period) nocturnal sleep duration, assessed by sleep diary | Baseline, End of Intervention (Day 77)
  Nocturnal sleep duration will be assessed by sleep diary
Change in average (over a 7-day period) 24-hour sleep duration, assessed by sleep diary | Baseline, End of Intervention (Day 77)
  24-hour sleep duration will be assessed by sleep diary
Change in average (over a 7-day period) sleep midpoint, assessed by sleep diary | Baseline, End of Intervention (Day 77)
  Sleep midpoint is the time half way between start and end of sleep, as assessed by sleep diary
Change in average (over a 7-day period) nocturnal sleep duration, assessed by activity tracker | Baseline, End of Intervention (Day 77)
  Nocturnal sleep duration will be assessed by activity tracker
Change in average (over a 7-day period) 24-hour sleep duration, assessed by activity tracker | Baseline, End of Intervention (Day 77)
  24-hour sleep duration will be assessed by activity tracker
Change in average (over a 7-day period) sleep efficiency, assessed by activity tracker | Baseline, End of Intervention (Day 77)
  Sleep Efficiency is the percentage of the sleep period spent asleep, as measured by activity tracker
Change in average (over a 7-day period) sleep midpoint, assessed by activity tracker | Baseline, End of Intervention (Day 77)
  Sleep midpoint is the time half way between start and end of sleep, as assessed by sleep diary

CONTACTS AND LOCATIONS:
Overall Officials: Christina Barkauskas, MD, Study Chair — Duke Clinical Research Institute; Susan Redline, MD MPH, Study Chair — Brigham and Women's Hospital
Locations (1):
- All sites listed under NCT06404086, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The summary of results will be shared on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT06404099/ICF_000.pdf